CLINICAL TRIAL: NCT00697671
Title: Pilot Study of Haploidentical Natural Killer Cell Infusions for Poor Prognosis Non-AML Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Assisi Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NKHEM
Record Dates: First submitted 2008-04-14; First posted 2008-06-16 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Acute Lymphoblastic Leukemia; Chronic Myelogenous Leukemia; Juvenile Myelomonocytic Leukemia; Myelodysplastic Syndrome; Non-Hodgkin's Lymphoma
Keywords: NK cell infusion; Immunotherapy; hematologic malignancy; Miltenyi Biotec device; haploidentical donor
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myelomonocytic, Juvenile; Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin; Hematologic Neoplasms | interventions — Immunotherapy; Interleukin-2; Clofarabine; Cyclophosphamide; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Strata A (Other): Patients with ALL, CML, JMML, MDS, or NHL with bone marrow relapse after stem cell transplant.
  Interventions: Other: NK Cell Infusion; Biological: Immunotherapy; Device: Miltenyi Biotec CliniMACS device; Drug: Interleukin-2 (IL-2); Drug: Clofarabine; Drug: Cyclophosphamide; Drug: Etoposide
- Strata B (Other): Patients with ALL, CML, JMML , MDS, or NHL with primary induction failure and persistent disease; or participants with relapsed ALL, CML, JMML, MDS, or NHL with persistent disease after re-induction
  Interventions: Other: NK Cell Infusion; Biological: Immunotherapy; Device: Miltenyi Biotec CliniMACS device; Drug: Interleukin-2 (IL-2); Drug: Clofarabine; Drug: Cyclophosphamide; Drug: Etoposide

INTERVENTIONS:
Other: NK Cell Infusion — All participants will receive a 4 day regimen of chemotherapy (clofarabine, cyclophosphamide, and etoposide) followed by an infusion of HLA partially matched family member donor NK cells processed through the use of the investigational CliniMACS device. Interleukin-2 (IL-2) will be given three times per week post-infusion for a minimum of 2 weeks. IL-2 administration will continue until donor NK cells are no longer detectable in the recipient, and, at that time, will be discontinued
Biological: Immunotherapy — All participants will receive a 4 day regimen of chemotherapy (clofarabine, cyclophosphamide, and etoposide) followed by an infusion of HLA partially matched family member donor NK cells processed through the use of the investigational CliniMACS device. Interleukin-2 (IL-2) will be given three times per week post-infusion for a minimum of 2 weeks. IL-2 administration will continue until donor NK cells are no longer detectable in the recipient, and, at that time, will be discontinued.
Device: Miltenyi Biotec CliniMACS device — All participants will receive a 4 day regimen of chemotherapy (clofarabine, cyclophosphamide, and etoposide) followed by an infusion of HLA partially matched family member donor NK cells processed through the use of the investigational CliniMACS device. Interleukin-2 (IL-2) will be given three times per week post-infusion for a minimum of 2 weeks. IL-2 administration will continue until donor NK cells are no longer detectable in the recipient, and, at that time, will be discontinued.
Drug: Interleukin-2 (IL-2) — All participants will receive a 4 day regimen of chemotherapy (clofarabine, cyclophosphamide, and etoposide) followed by an infusion of HLA partially matched family member donor NK cells processed through the use of the investigational CliniMACS device. Interleukin-2 (IL-2) will be given three times per week post-infusion for a minimum of 2 weeks. IL-2 administration will continue until donor NK cells are no longer detectable in the recipient, and, at that time, will be discontinued.
Drug: Clofarabine — All participants will receive a 4 day regimen of chemotherapy (clofarabine, cyclophosphamide, and etoposide) followed by an infusion of HLA partially matched family member donor NK cells processed through the use of the investigational CliniMACS device. Interleukin-2 (IL-2) will be given three times per week post-infusion for a minimum of 2 weeks. IL-2 administration will continue until donor NK cells are no longer detectable in the recipient, and, at that time, will be discontinued.
Drug: Cyclophosphamide — All participants will receive a 4 day regimen of chemotherapy (clofarabine, cyclophosphamide, and etoposide) followed by an infusion of HLA partially matched family member donor NK cells processed through the use of the investigational CliniMACS device. Interleukin-2 (IL-2) will be given three times per week post-infusion for a minimum of 2 weeks. IL-2 administration will continue until donor NK cells are no longer detectable in the recipient, and, at that time, will be discontinued.
Drug: Etoposide — All participants will receive a 4 day regimen of chemotherapy (clofarabine, cyclophosphamide, and etoposide) followed by an infusion of HLA partially matched family member donor NK cells processed through the use of the investigational CliniMACS device. Interleukin-2 (IL-2) will be given three times per week post-infusion for a minimum of 2 weeks. IL-2 administration will continue until donor NK cells are no longer detectable in the recipient, and, at that time, will be discontinued.

SUMMARY:
The prognosis of pediatric patients with hematologic malignancies whose disease is primarily refractory or those who experience a chemotherapy resistant bone marrow relapse is extremely poor. When new agents or chemotherapeutic regimens are unable to induce remission in this patient population, hematopoietic stem cell transplant (HSCT) is also a poor alternative. Thus, in this very high risk group, additional attempts at remission induction with various combinations of chemotherapy alone will unlikely improve outcome and will contribute to overall toxicity. Alternative therapies are needed in these patients with chemotherapy resistant disease.

Immunotherapy with natural killer (NK) cell infusion has the potential to decrease toxicity and induce hematologic remission. NK cells can kill target cells, including leukemia cells, without prior exposure to those cells. In patients undergoing allogeneic HSCT, several studies have demonstrated the powerful effect of NK cells against leukemia. Furthermore, NK cell infusions in patients with primary refractory or multiple-relapsed leukemia have been shown to be well tolerated and void of graft-versus-host disease effects. In this high risk group, complete leukemic remission has been observed in several of these patients after NK cell infusion.

With the current technology available at St. Jude, we have developed a procedure to purify NK cells from adult donors. This protocol will assess the safety of chemotherapy and IL-2 administration to facilitate transient NK-cell engraftment in research participants who have chemotherapy refractory hematologic malignancies including acute lymphoblastic leukemia, chronic myelogenous leukemia, juvenile myelomonocytic leukemia, myelodysplastic syndrome, or non-Hodgkin's lymphoma. In this same cohort, we will also intend to explore the efficacy of NK cells infused in those participants who have chemotherapy refractory disease.

DETAILED DESCRIPTION:
This study will evaluate the persistence, phenotype and function of donor NK cells as well as exploring the efficacy of the infusion in research participants with chemotherapy refractory hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* At least two weeks since receipt of last biological therapy, chemotherapy, or radiation therapy.
* Has a suitable adult family member donor available for NK cell donation.
* No current pleural or pericardial effusion.
* HIV negative
* Adequate clinical standing as evidenced by being within multiple renal, hepatic, pulmonary, and neurological required testing parameters.

Exclusion Criteria:

* Pregnant or lactating

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2007-03; Primary Completion 2013-02 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
To assess the safety of chemotherapy and IL-2 administration to facilitate transient NK-cell engraftment in research participants with chemotherapy refractory non-acute myelogenous leukemia (non-AML) hematologic malignancies | 4 months post infusion

SECONDARY OUTCOMES:
To study the persistence, phenotype and function of donor natural killer (NK) cells after infusion in research participants with chemotherapy refractory hematologic malignancies. | 4 months infusion
To explore the efficacy of NK cell infusion in research participants with chemotherapy refractory hematologic malignancies | 4 months infusion

CONTACTS AND LOCATIONS:
Overall Officials: Wing Leung, MD, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org